CLINICAL TRIAL: NCT01416116
Title: Tolerability of QUTENZATM When Applied After Pre-treatment With Lidocaine or Tramadol in Subjects With Peripheral Neuropathic Pain - A Randomized, Multi-center, Assessor-blinded Study
Brief Title: Method of Pre-treatment for Application of QUTENZA Capsaicin 8% Patch
Acronym: LIFT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QTZ-EC-0002; 2010-023258-34 (EudraCT Number)
Record Dates: First submitted 2011-08-11; First posted 2011-08-12 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: or Peripheral Nerve Injury (PNI); Peripheral Neuropathic Pain (PNP) Due to Postherpetic Neuralgia (PHN)
Keywords: Tramadol; QUTENZA; Pre-treatment; Tolerability
MeSH Terms: conditions — Peripheral Nerve Injuries | interventions — Capsaicin; Transdermal Patch; Lidocaine; Tramadol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tramadol (Experimental): Tramadol prior to QUTENZA
  Interventions: Drug: QUTENZA; Drug: Tramadol
- Lidocaine (Experimental): Lidocaine prior to QUTENZA
  Interventions: Drug: QUTENZA; Drug: Lidocaine

INTERVENTIONS:
Drug: QUTENZA — topical
  Other Names: capsaicin 8% patch
Drug: Lidocaine — topical
  Arms: Lidocaine
Drug: Tramadol — oral
  Arms: Tramadol

SUMMARY:
The Summary of product characteristics (SmPC) for QUTENZA advises that topical anaesthetic is applied prior to the application of QUTENZA. This is a multi-center, randomized, assessor-blinded study which will investigate the use of an oral analgesic as an alternative form of pre-treatment for QUTENZA.

DETAILED DESCRIPTION:
All patients will be treated with QUTENZA for 60 minutes. Patients will be randomized to one of two arms- application of topical anaesthetic (lidocaine cream) or an oral analgesic (tramadol oral tables) prior to application of QUTENZA. Patients will be followed up for 7 days to monitor pain scores and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of postherpetic neuralgia or neuropathic pain due to peripheral nerve injury
* Daily pain score ≥ 4 for average pain both at the Screening Visit and at the Treatment Visit
* Intact, non-irritated, dry skin over the painful area(s) to be treated

Exclusion Criteria:

* Significant ongoing or recurrent pain other than due to PHN or peripheral nerve injury
* Past or current history of Type I or Type II diabetes mellitus
* Active malignancy or treatment for malignancy within a year prior to the Treatment Visit

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2011-07-06 (Actual); Primary Completion 2012-04-25 (Actual); Study Completion 2012-04-25 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects who tolerate QUTENZA treatment | 60 minute application period
  A QUTENZA tolerant subject is defined as a subject receiving at least 90% of the intended patch duration.

SECONDARY OUTCOMES:
Duration of patch application | 60 minutes
Change in pain scores from baseline to subsequent timepoints on the day of patch application | 5, 25, 55, 85, 115 minutes on day of application and once a day on days 1, 2, 3
Proportion of subjects using pain medications and dose of pain medication(s) administered | day 1-5
Subject rated tolerability score | Baseline to end of study visit, day 7

CONTACTS AND LOCATIONS:
Overall Officials: Senior Study Manager, Late Phase Clinical Development & Operations, Study Director — Astellas Pharma Europe Limited
Locations (20):
- Belgium (3):
  - Site 102, Antwerp
  - Site 103, Genk
  - Site 101, Roeselare
- Czechia (3):
  - Site 202, Hradec Králové
  - Site 203, Olomouc
  - Site 201, Prague
- Denmark (2):
  - Site 302, Aalborg
  - Site 301, Aarhus
- Ireland (4):
  - Site 402, Cork
  - Site 403, Galway
  - Site 404, Galway
  - Site 401, Limerick
- Norway (2):
  - Site 502, Hamar
  - Site 501, Skien
- Slovakia (2):
  - Site 603, Košice
  - Site 602, Martin
- United Kingdom (4):
  - Site 702, Glasgow
  - Site 701, Liverpool
  - Site 704, Manchester
  - Site 703, Solihull

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=82